CLINICAL TRIAL: NCT03692754
Title: A Single-center Prospective Randomized Study of Atorvastatin in the Treatment of Newly Diagnosed Primary Immune Thrombocytopenia (ITP)
Brief Title: Atorvastatin in Management of Newly Diagnosed ITP
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Ming Hou, Professor and Director, Shandong University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Atorvastatin in ITP
Record Dates: First submitted 2018-09-29; First posted 2018-10-02 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-08

CONDITIONS: Immune Thrombocytopenia; Purpura, Thrombocytopenic
Keywords: Immune Thrombocytopenia
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic; Purpura, Thrombocytopenic | interventions — Atorvastatin; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- AT with 10 mg/d (Active Comparator): The patients will be given receive atorvastatin in 10 mg/d for 1 month plus dexamethasone 40mg/d for 4 days.
  Interventions: Drug: Atorvastatin 10mg; Drug: Dexamethasone
- AT with 20 mg/d (Active Comparator): The patients will be given atorvastatin in 20 mg/d for 1 month plus dexamethasone 40mg/d for 4 days.
  Interventions: Drug: Atorvastatin 20mg; Drug: Dexamethasone
- Dexamethasone (Experimental): The patients will be given dexamethasone 40mg/d for 4 days.
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Atorvastatin 20mg — Atorvastatin will be given in 20 mg po qn for 1 month
  Other Names: atorvastatin calcium
  Arms: AT with 20 mg/d
Drug: Atorvastatin 10mg — Atorvastatin will be given in 10 mg po qn for 1 month
  Other Names: atorvastatin calcium
  Arms: AT with 10 mg/d
Drug: Dexamethasone — Dexamethasone will be given in 40mg po qd for 4 days

SUMMARY:
The project was undertaking by Qilu Hospital of Shandong University in China. In order to report the efficacy and safety of atorvastatin for the treatment of adults with immune thrombocytopenia (ITP).

DETAILED DESCRIPTION:
The investigators anticipate to undertaking a parallel group, single-centre, randomised controlled trial of 30 ITP adult patients, which have no indications of glucocorticoid therapy (platelets count > 30*10^9/L )from Qilu Hospital of Shandong University in China.15 of the participants are randomly selected to receive atorvastatin in 20 mg/d combining with 10 mg/d for 6 months. Platelet count, bleeding and other symptoms were evaluated before and after treatment, adverse events are also recorded throughout the study in order to report the efficacy and safety of atorvastatin for the treatment of adults with ITP.

ELIGIBILITY:
Inclusion Criteria:

1. Meet the diagnostic criteria for immune thrombocytopenia.
2. within 3 months from diagnosis,untreated patients, may be male orfemale, between the ages of 18 ~ 80 years.
3. To show a platelet count > 30×10^9/L and without bleeding manifestations.

Exclusion Criteria:

1. Received chemotherapy or anticoagulants or other drugs affecting theplatelet counts within 3 months before the screening visit.
2. Received steroids or other effective therapy for immune thrombocytopenia.
3. Current HIV infection or hepatitis B virus or hepatitis C virus infections.
4. Severe medical condition (lung, hepatic or renal disorder) other than ITP.
5. Unstable or uncontrolled disease or condition related to or impacting cardiac function (e.g., unstable angina, congestive heart failure, uncontrolled hypertension or cardiac arrhythmia)
6. Female patients who are nursing or pregnant, who may be pregnant, or who contemplate pregnancy during the study period.
7. Have a known diagnosis of other autoimmune diseases, established in the medical history and laboratory findings with positive results for the determination of antinuclear antibodies, anti-cardiolipin antibodies, lupus anticoagulant or direct Coombs test.
8. Patients who are deemed unsuitable for the study by the investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-11-01 (Estimated); Primary Completion 2021-12-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of platelet response | up to 1 year per subject
  Platelet count will be observed at 1 month, 3 months, 6 months and 12 months after atorvastatin therapy

SECONDARY OUTCOMES:
Therapy associated adverse events | up to 1 year per subject
  The number and frequency of therapy associated adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Ming Hou, Dr, Principal Investigator — Shandong University
Locations (1):
- Qilu hospital, Shandong University, Jinan, Shandong, China